CLINICAL TRIAL: NCT07128693
Title: A Single-center, Multicohort, Phase II Clinical Study Evaluating the Combination Therapy of Sacituzumab Tirumotecan in Patients With Unresectable, Locally Advanced, Recurrent, or Metastatic Esophageal Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Feng Wang, Professor, The First Affiliated Hospital of Zhengzhou University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-KY-0942
Record Dates: First submitted 2025-08-14; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — tislelizumab; anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First-line treatment with Sacituzumab Tirumotecan in combination with tislelizumab (Experimental): First-line treatment with Sacituzumab Tirumotecan in combination with tislelizumab
  Interventions: Drug: Sacituzumab Tirumotecan in combination with tislelizumab
- Second-line treatment with Sacituzumab Tirumotecan in combination with anlotinib (Experimental): Second-line treatment with Sacituzumab Tirumotecan in combination with anlotinib
  Interventions: Drug: Sacituzumab Tirumotecan in combination with anlotinib

INTERVENTIONS:
Drug: Sacituzumab Tirumotecan in combination with tislelizumab — Sacituzumab Tirumotecan 5mg/kg, iv, d1, Q2W ,until disease progression or intolerable toxicity.
  Tislelizumab，200 mg, iv, d1, Q3W, until disease progression or intolerable toxicity.
  Arms: First-line treatment with Sacituzumab Tirumotecan in combination with tislelizumab
Drug: Sacituzumab Tirumotecan in combination with anlotinib — Sacituzumab Tirumotecan 5mg/kg, iv, d1, Q2W ,until disease progression or intolerable toxicity.
  Anlotinib 12mg QD po d1-14，Q3W,until disease progression or intolerable toxicity.
  Arms: Second-line treatment with Sacituzumab Tirumotecan in combination with anlotinib

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of the combined treatment with Sacituzumab Tirumotecan in patients with unresectable locally advanced/recurrent or metastatic esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of informed consent signing.
2. Diagnosed as unresectable locally advanced/recurrent or metastatic esophageal squamous cell carcinoma by histology/pathology.
3. Cohort 1: Have never received any anti-tumor systemic treatment before, including but not limited to immunotherapy, targeted therapy, chemotherapy, etc. Cohort 2: Patients who have experienced progression or intolerance after receiving first-line systemic chemotherapy or chemotherapy combined with immunotherapy (which may include regimens based on platinum, taxanes or fluorouracil) (patients with progression after maintenance treatment following first-line chemotherapy can also be included).
4. For patients with brain metastases, those who are asymptomatic or have stable symptoms of brain metastases are eligible for enrollment.
5. The provision of tissue specimens is not mandatory. Patients can still be enrolled if there is no tissue specimen available.
6. According to RECIST v1.1, the investigator should assess that there is at least one measurable target lesion that has not been irradiated.
7. ECOG performance status score of 0 or 1.
8. Expected survival time ≥ 12 weeks.
9. Adequate organ and bone marrow function(with no receipt of blood transfusions, recombinant human thrombopoietin, or colony-stimulating factors within two weeks prior to first drug administration), defined as follows:

   1. Blood routine: Neutrophil count (NEUT#) ≥ 1.5×109/L; Platelet (PLT) ≥100×109/L; Hemoglobin ≥ 90g/L.
   2. Liver function: Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 2.5 times the upper limit of normal (ULN); total bilirubin (TBIL) ≤ 1.5 times ULN;
   3. Renal function: Ccr ≥ 60 ml/min (Cockcroft-Gault formula provided).
   4. International Normalized Ratio (INR), activated partial thromboplastin time (APTT), and prothrombin time (PT) values are ≤ 1.5 times the upper limit of normal (ULN).
10. For female subjects of childbearing potential and male subjects with reproductive potential, a commitment to effective medical contraception is required from the date of informed consent signing through 6 months after the last dose administration.
11. The subjects voluntarily joined this study, signed the informed consent form, and were able to comply with the visit and related procedures as stipulated in the protocol.

Exclusion Criteria:

1. Having participated in other drug clinical trials within 4 weeks before enrollment.
2. Cohort 1: Having previously received treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibodies, or any other antibodies or drugs specifically targeting T-cell co-stimulation or checkpoint pathways.
3. Cohort 2: Having previously received anlotinib or other anti-angiogenic drugs; patients with tumor invasion of large blood vessels shown by imaging, or those judged to be highly likely to have tumors invading important blood vessels during the subsequent study period, leading to fatal massive bleeding; patients with bleeding tendencies such as acute gastrointestinal bleeding, persistent bleeding disorders, or coagulation dysfunction.
4. Patients with multiple factors affecting oral drug administration (such as inability to swallow, post-gastrointestinal resection, chronic diarrhea, intestinal obstruction, etc.).
5. Prior treatment with TROP2-targeted therapy and/or topoisomerase I inhibitors.
6. A history of other malignant tumors within the past 5 years, excluding cured cervical carcinoma in situ, basal cell carcinoma, or squamous cell carcinoma of the skin.
7. Known history of allergy to the drugs in this protocol and their components.
8. Positive for human immunodeficiency virus (HIV) test or history of acquired immunodeficiency syndrome (AIDS); known active syphilis infection.
9. History of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
10. Vaccinated with live vaccine within 30 days before the first study drug administration.
11. 7.A history of interstitial lung disease (ILD) or non-infectious pneumonia requiring corticosteroid therapy, or current ILD or non-infectious pneumonia, or suspected ILD or non-infectious pneumonia at screening that cannot be ruled out by imaging; clinically significant pulmonary impairment due to concurrent lung conditions, including but not limited to underlying pulmonary disorders (e.g., pulmonary embolism within 3 months prior to study entry, severe asthma, severe chronic obstructive pulmonary disease [COPD], restrictive lung disease, pleural effusion), autoimmune, connective tissue, or inflammatory disorders with potential pulmonary involvement (e.g., rheumatoid arthritis, Sjogren's syndrome, sarcoidosis), or prior pneumonectomy.
12. Active autoimmune diseases requiring systemic therapy within the past two years (hormone replacement therapy is excluded from systemic treatment, including conditions such as type 1 diabetes, hypothyroidism managed with thyroid hormone replacement alone, and adrenal or pituitary insufficiency treated solely with physiological doses of glucocorticoid replacement therapy).
13. Active infections requiring systemic treatment within 2 weeks prior to the first dose administration.
14. Concomitant diseases that, in the investigator's judgment, pose a significant risk to patient safety or may interfere with study completion, including but not limited to medication-uncontrolled hypertension, severe diabetes, or active infections.
15. A documented history of severe dry eye syndrome, severe meibomian gland dysfunction and/or blepharitis, or corneal disorders associated with delayed corneal healing.
16. Female patients who are pregnant, lactating, or of childbearing potential with a positive baseline pregnancy test; female patients of childbearing age who are unwilling to adopt effective contraceptive measures during the treatment with the study drug and within 6 months after the last dose.
17. Any other circumstances deemed by the investigator to make the patient unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
PFS | Up to 24 months
  PFS is defined as the time from the first administration to the first documented progressive disease (PD) per RECIST 1.1 by investigators or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
ORR | Up to 24 months
  ORR is defined as the percentage of participants with Complete Response or Partial Response per RECIST 1.1 assessed by the investigators.
DCR | Up to 24 months
  DCR is defined as the proportion of subjects with complete response (CR), partial response (PR) and stable disease (SD) among all subjects.
DOR | Up to 24 months
  DOR is defined as the time interval from the first documented disease response to disease progression or death (whichever occurs first)
OS | Up to 24 months
  OS is defined as the time from the first receipt of treatment under the study protocol to the death of the subject due to any reason.
Adverse Events (AEs) | Up to 24 months
  The number of participants experiencing an AE will be assessed